CLINICAL TRIAL: NCT02109705
Title: Porphyromonas Gingivalis - a Responsible Pathogen in Alzheimer's Disease?
Brief Title: Porphyromonas Gingivalis and Alzheimer's Disease
Acronym: PGNEURO
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: PG001
Record Dates: First submitted 2014-03-31; First posted 2014-04-10 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2014-12

CONDITIONS: Alzheimer's Disease; Dementia; Periodontitis
MeSH Terms: conditions — Alzheimer Disease; Dementia; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — GCF, Liquor, Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Alzheimer's Disease
- other Dementia
- cognitive healthy

SUMMARY:
With this study the investigators would like to analyze the the role of periodontal disease and especially the role of Porphyromonas gingivalis in initiation and progression of Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* age 40-70
* caucasian origin
* dementia (Alzheimer's or other dementia)
* cognitive healthy (need for spinal anesthesia)

Exclusion Criteria:

* use of antibiotics within las 6 months
* pregnancy
* another illness explaining the symptoms in a better way
* smoking (>10 cigarettes)
* patients who have a legal custodian

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 Patients with Dementia (30 with Alzheimer's and 30 with another Dementia) 30 cognitive healthy patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Cmax Antibody Levels against Gingipains | Baseline
  laboratory analysis

SECONDARY OUTCOMES:
Cmax Beta-Amyloid | Baseline
  laboratory analysis

OTHER OUTCOMES:
Cmax: Periodontal pathogens | Baseline
  laboratory analysis
U enzyme activities | Baseline
  laboratory analysis
Cmax: inflammatory cytokines | Baseline
  laboratory analysis

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Laugisch, Dr med dent MAS, Principal Investigator — Department of Periodontology
Locations (1):
- Department of Periodontology, Münster, Germany